CLINICAL TRIAL: NCT03695328
Title: Effect of Nutrition and Physical Activity on Bone Status in 6-12 Years Children
Brief Title: Physical Activity, Dietary Intake and Bone Status in 6-12 Years Children
Acronym: Nutri-Bone
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, KAMBAS ANTONIS, Professor, Democritus University of Thrace
Other Study IDs: Nutri-Bone DUTH
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Bone Status
MeSH Terms: interventions — Eating

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- physical activity level: Children categorized either in the group with moderate to vigorous physical activity or in the group with low physical activity according the accelerometer's measures
  Interventions: Behavioral: physical activity level
- dietary intake: Childrens' 24th dietary recalls for 7 days analyzed for protein, calcium, vitamin D and phosphorus intake and they categorized according the RDAs above or below them.
  Interventions: Behavioral: Dietary Intake

INTERVENTIONS:
Behavioral: physical activity level
  Groups: physical activity level
Behavioral: Dietary Intake
  Groups: dietary intake

SUMMARY:
Peak bone mass acquisition through childhood and adolescence has been associated with lower risk of osteopenia and osteoporosis in the elderly. The main factors that influence bone mass are the non-modifiable, such as genetics, ethnicity and sex, and the modifiable ones which are nutrition and physical activity or exercise. In the literature are references that demonstrates positive effects of high physical activity, adequate intakes of macro- and micronutrients on bone mass both in adults and in children. Bone mineralization is more adaptive in childrens' growing bones and this is an opportunity for stronger effects by mechanical stimuli during physical activity. The presence of a diet complete of nutrient intakes seems to strengthen the effects of mechanical loads on bone growth and mineralization. The present trial aimed to evaluate the effects of physical activity and nutrition intakes on bone mass in pre-pubertal children.

DETAILED DESCRIPTION:
The sample of this study was healthy pre-pubertal boys and girls (N=210) who had training age 0-1 years. Data collection included anthropometric measurements, blood sampling, body composition, bone measurements and physical performance measurements. Nutritional intake was recorded for seven consecutive days in order to evaluate nutrient intakes using an appropriate software and habitual physical activity was measured for the same days using accelerometers. Pubertal stage determined by Tanner scale. All measurements were made only once at the beginning of school year.

ELIGIBILITY:
Inclusion Criteria:

* were 6-12 years and pre-pubertal
* were healthy and had no prior bone fractures or related surgical operation
* their body fat was <30%, e) had no history of growth irregularities
* were not receiving agents or drugs that affect bone tissue (e.g. Gonadotropin-Releasing Hormone (GnRH) agonists, antiresorptive, bisphosphonates, etc.)

Exclusion Criteria:

* had prior bone fractures or related surgical operation
* their body fat was >30%
* had history of growth irregularities
* were receiving agents or drugs that affect bone tissue (e.g. GnRH agonists, antiresorptive, bisphosphonates, etc.)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary schoolchildren (boys and girls) aged 6-12 years and were at pre-pubertal stage.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2015-10-25 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Whole body bone mineral density | 1 day (Once)
  Measured by Dual-X-ray Absoroptiometry
Lumbar spine bone mineral density | 1 day (Once)
  Measured by Dual-X-ray Absoroptiometry
Hips bone mineral density | 1 day (Once)
  Measured by Dual-X-ray Absoroptiometry
Whole body mineral content | 1 day (Once)
  Measured by Dual-X-ray Absoroptiometry
Lumbar spine bone mineral content | 1 day (Once)
  Measured by Dual-X-ray Absoroptiometry
Hips bone mineral content | 1 day (Once)
  Measured by Dual-X-ray Absoroptiometry
Body composition | 1 day (Once)
  Measured by Dual-X-ray Absoroptiometry and skinfolds
Muscular strength | 1 day (Once)
  Handgrip strength
Cardiovascular endurance | 1 day (Once)
  20m shuttle run test
Flexibility | 1 day (Once)
  Sit and reach test

SECONDARY OUTCOMES:
Sclerostin | 1 day (Once)
  Measured in blood samples with an appropriate kit
Serum vitamin D | 1 day (Once)
  Measured in blood smaples
Serum calcium | 1 day (Once)
  Measured in blood smaples
Pubertal Stage | 1 day (Once)
  Evaluated with Tanner Stage protocol

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Stampoulis, PhD student, Principal Investigator — Democritus University of Thrace, Department of Physical Education & Sports Sciencies